CLINICAL TRIAL: NCT04460339
Title: Changes in Body Core Temperature During a 25-km Open Water Race in Elite Swimmers: Identifying Predictors for Hypothermia and Dropouts
Brief Title: Thermoregulation During a 25-km Open Water Race
Acronym: THERMO25
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: THERMO25
Record Dates: First submitted 2020-06-27; First posted 2020-07-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2020-07

CONDITIONS: Hypothermia Due to Cold Environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Swimming participants in the 25-km — The 25-km race was the French national Open Championship event and participants were the swimmers registered for the race who volunteered to participate in this study

SUMMARY:
Open water swimming is a swimming discipline which takes place in outdoor water such as open oceans, lakes, and rivers. Elite swimmers are exposed to hypothermia when swimming in cold water, especially in long duration races, such as the 25-km race. The objective of this study is to evaluate the change in body core temperature in swimmers with continuous temperature monitoring during a 25-km race. The secondary objective is to identify the predictors of hypothermia and hypothermia-related drop-out.

ELIGIBILITY:
Inclusion Criteria:

* competitors of the 25-km French Open Water Championship
* participants who volunteered for this study
* written consent was obtained from all participants, as well as their legal representatives when applicable (i.e. parents for under age participants).

Exclusion Criteria:

* swallowing disorders
* transit disorders
* MRI scheduled within 48 hours

Ages: 15 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: All the competitors of the 25-km French Open Water Championship who volunteered for this study
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-26 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Change in Body Core Temperature | Continuous measurement was collected from 30 minutes before the race until 2 hours after the end of the race for each swimmer
  Measurement of Body Core Temperature using an ingestible electronic sensor (e-Celsius®, BodyCap , Caen, France) which provide a continuous validated measurement
Change in Water Temperature | Continuous measurement was collected from 30 minutes before the race until 2 hours after the end of the race for each swimmer
  Measurement of the Water Temperature using an electronic sensor (iButton® Maxim Integrated) which provide a continuous validated measurement

SECONDARY OUTCOMES:
Body composition, body mass | One measurement assessed the day before the race
  Body mass (in kg) was measured using bioelectrical impedance analysis (mBCA 525, Seca, Germany).
Body composition, fat mass | One measurement assessed the day before the race
  Fat mass (in kg, % of body mass [fat mass and body mass were combined to report % of body mass) was measured using bioelectrical impedance analysis (mBCA 525, Seca, Germany).
Body composition, fat-free mass | One measurement assessed the day before the race
  Fat-free mass (in kg, % of body mass [fat-free mass and body mass were combined to report % of body mass) was measured using bioelectrical impedance analysis (mBCA 525, Seca, Germany).
Body composition, muscle mass | One measurement assessed the day before the race
  Muscle mass (in kg, % of body mass [muscle mass and body mass were combined to report % of body mass) was measured using bioelectrical impedance analysis (mBCA 525, Seca, Germany).
Perception of Cold | One measurement assessed immediately at the end of the race
  Immediately at the end of the race participants' perception of cold was assessed using the Cold Discomfort Scale (CDS, with rating from 0-to-10 over 10, where 0 indicates no experience of cold and 10 indicates unbearable cold)
Performance | Time at each lap of 2500m and at the end of the race
  Time at each lap and swimming race timing was collected using the official swimming timing from the race organisers and French Federation
Dropout rate | During the swimming race and data were collected immediately after dropout for each swimmer who dropped out
  Swimmers who dropout were identified and cause for dropout was collected

CONTACTS AND LOCATIONS:
Overall Officials: Joffrey Drigny, MD MSC, Principal Investigator — CHU Caen Normandie
Locations (1):
- CHU Caen Normandie, Caen, France